CLINICAL TRIAL: NCT02217592
Title: Causes and Factors Associated With Outcomes in Community-acquired Sepsis and Severe Sepsis in Northeast (NE) Thailand
Brief Title: Causes and Factors Associated With Outcomes in Community-acquired Sepsis and Severe Sepsis in Northeast Thailand
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other); National Institutes of Health (NIH) (NIH); University of Washington (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: MICRO1206; 1R01HL113382 (NIH)
Record Dates: First submitted 2014-08-01; First posted 2014-08-15 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Sepsis; Severe Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood. Urine, pus, sputum, throat swab, and stool (if available)
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study to identify the aetiology and factors associated with outcome of community-acquired sepsis and severe sepsis in Northeast Thailand.

Potential study participants will be adult patients who are presented at the hospital with community-acquired sepsis. Clinical specimens (including blood, urine, sputum and throat swabs) will be collected from each participant on admission for culture, PCR and serological tests, and other laboratory tests, including inflammatory markers and genotyping. Participants' treatment will be closely monitored during the duration of their hospital stay. Blood will be again collected at 72 hours after admission. Participants will be contacted at 28 days after admission to determine clinical outcome by phone interview with standardized script.

There will be a total of 5,020 patients enrolled in this study over 3 years.

DETAILED DESCRIPTION:
Primary objective: To determine the causes of community-acquired sepsis and severe sepsis in NE Thailand.

Secondary Objectives:

1. To define the clinical outcome of community-acquired sepsis and severe sepsis in NE Thailand.
2. To determine factors associated with inflammatory response, organ failure, and mortality in community-acquired sepsis and severe sepsis in NE Thailand, including causes of sepsis, sepsis resuscitation, antimicrobial treatment and genetic factors.
3. To evaluate diagnostic tests for infection in community-acquired sepsis and severe sepsis in NE Thailand.

NOTE: THIS STUDY IS CO-SPONSORED BY

1. University of Oxford
2. University of Washington

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years old
* Thai nationality
* Required hospitalization as decided by the attending physician
* Documented by attending physician that an infection is the primary cause of illness leading to the hospitalization. These can be infections due to any pathogens (bacteria, viruses, fungi and parasites)
* Presence of any 3 of the following Systemic Inflammatory Response Syndrome (SIRS)

  * Fever or hypothermia (Core body temperature defined as > 38.3 C or < 36.0 C)
  * Tachycardia (heart rate > 90 beats per minute)
  * Tachypnea (respiratory rate > 20 per minute)
  * Arterial hypotension (systolic blood pressure (SBP) < 90 mmHg, mean arterial pressure (MAP) < 70 mmHg, or SBP decrease > 40 mmHg)
  * White blood cell (WBC) > 12,000/µL < 4000/µL or immature forms > 10%
  * Platelet count < 100,000/microlitre
  * Altered mental status with Glasgow Coma Score (GCS) < 15
  * Hypoxemia (Pulse Oximetry Level < 95)
  * Ileus
  * Significant edema or positive fluid balance
  * Decreased capillary refill or mottling
  * Hyperglycemia (plasma glucose > 140 mg/dL) in the absence of diabetes
  * Plasma C-reactive protein > 2 SD above the normal value
  * Plasma procalcitonin > 2 SD above the normal value
  * Arterial hypoxemia (PaO2 / FIO2 < 300)
  * Acute oliguria (urine output < 0.5 mL/kg/hr or 45 mmol/L for 2 hours)
  * Creatinine increase > 0.5 mg/dL
  * INR > 1.5 or aPTT > 60 seconds
  * Plasma total bilirubin > 4 mg/dl or 70 mmol/L
  * Hyperlactatemia (> 1 mmol/L)

Exclusion Criteria

* Infection is not suspected to be a primary cause of the current illness episode leading to the hospitalization. For example, community-acquired sepsis or severe sepsis is considered to be due to stroke, cardiovascular diseases, acute myocardial infarction, cancer, burn, injury, and trauma
* Hospitalized at this study site for this current episode for more than 24 hours before enrollment
* Hospitalized for this current episode for more than 72 hours at another primary/referring hospital
* Prior to this current episode, the patient was admitted to any hospital within the last 30 days
* Prior to enrolment, it is documented by the attending physician that hospital acquired infection is associated with the cause of sepsis or severe sepsis

Please note that the following conditions are not exclusion criteria, and patients with the following conditions can be enrolled into the study

* Confirmed diagnosis by any method of an infection as a major cause of illnesses leading to hospitalization. For example, a patient who already has had a definite diagnosis of malarial infection by blood smear
* Clinical diagnosis of any specific disease or any specific syndromes such as acute infective diarrhea, acute pneumonia, acute encephalomyelitis and acute myocarditis
* Suspected of having both infectious and non-infectious diseases and infectious disease is a primary cause of illnesses (primary diagnosis) leading to the hospitalization. For example, acute pneumonia with stroke as an underlying disease, etc
* Patients who are admitted to other hospitals and referred to the study site. For example a referred patient who admit to the first hospital less than 48 hours prior to enrollment
* Patients fulfilling the inclusion criteria without having result of complete blood count or result of all parameters in the inclusion criteria. For example, a patient who has hypothermia, tachycardia and tachypnea completes the criteria of SIRS even without the result of complete blood count or the result of other parameters such as INR, or plasma procalcitonin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients, 18 years old with community-acquired sepsis or severe sepsis in Northeast Thailand
Sampling Method: Probability Sample
Enrollment: 5020 (Actual)
Dates: Start 2012-05-20 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage of enrolled subjects specified by bacterial/viral infection | 3 Years

SECONDARY OUTCOMES:
Percentage of deaths caused by community-acquired sepsis and severe sepsis in Northeast Thailand | 3 Years
Sensitivities and specificities of diagnostic tests for infection in community-acquired sepsis and severe sepsis in Northeast Thailand | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Direk Limmathurotsakul, Principal Investigator — Mahidol-Oxford Tropical Medicine Research Unit (MORU), Faculty of Tropical Medicine, Mahidol university, Thailand
Locations (1):
- Sappasithiprasong Hospital, Ubon Ratchathani, Thailand

REFERENCES:
- [Background] Limmathurotsakul D, Wuthiekanun V, Chantratita N, Wongsuvan G, Amornchai P, Day NP, Peacock SJ. Burkholderia pseudomallei is spatially distributed in soil in northeast Thailand. PLoS Negl Trop Dis. 2010 Jun 1;4(6):e694. doi: 10.1371/journal.pntd.0000694. PMID 20532233
- [Background] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Background] Cheng AC, West TE, Limmathurotsakul D, Peacock SJ. Strategies to reduce mortality from bacterial sepsis in adults in developing countries. PLoS Med. 2008 Aug 19;5(8):e175. doi: 10.1371/journal.pmed.0050175. PMID 18752342
- [Background] Maitland K, Kiguli S, Opoka RO, Engoru C, Olupot-Olupot P, Akech SO, Nyeko R, Mtove G, Reyburn H, Lang T, Brent B, Evans JA, Tibenderana JK, Crawley J, Russell EC, Levin M, Babiker AG, Gibb DM; FEAST Trial Group. Mortality after fluid bolus in African children with severe infection. N Engl J Med. 2011 Jun 30;364(26):2483-95. doi: 10.1056/NEJMoa1101549. Epub 2011 May 26. PMID 21615299
- [Background] Suttinont C, Losuwanaluk K, Niwatayakul K, Hoontrakul S, Intaranongpai W, Silpasakorn S, Suwancharoen D, Panlar P, Saisongkorh W, Rolain JM, Raoult D, Suputtamongkol Y. Causes of acute, undifferentiated, febrile illness in rural Thailand: results of a prospective observational study. Ann Trop Med Parasitol. 2006 Jun;100(4):363-70. doi: 10.1179/136485906X112158. PMID 16762116
- [Background] Gasem MH, Wagenaar JF, Goris MG, Adi MS, Isbandrio BB, Hartskeerl RA, Rolain JM, Raoult D, van Gorp EC. Murine typhus and leptospirosis as causes of acute undifferentiated fever, Indonesia. Emerg Infect Dis. 2009 Jun;15(6):975-7. doi: 10.3201/eid1506.081405. PMID 19523308
- [Background] Phongmany S, Rolain JM, Phetsouvanh R, Blacksell SD, Soukkhaseum V, Rasachack B, Phiasakha K, Soukkhaseum S, Frichithavong K, Chu V, Keolouangkhot V, Martinez-Aussel B, Chang K, Darasavath C, Rattanavong O, Sisouphone S, Mayxay M, Vidamaly S, Parola P, Thammavong C, Heuangvongsy M, Syhavong B, Raoult D, White NJ, Newton PN. Rickettsial infections and fever, Vientiane, Laos. Emerg Infect Dis. 2006 Feb;12(2):256-62. doi: 10.3201/eid1202.050900. PMID 16494751
- [Background] Wijedoru LP, Kumar V, Chanpheaktra N, Chheng K, Smits HL, Pastoor R, Nga TV, Baker S, Wuthiekanun V, Peacock SJ, Putchhat H, Parry CM. Typhoid fever among hospitalized febrile children in Siem Reap, Cambodia. J Trop Pediatr. 2012 Feb;58(1):68-70. doi: 10.1093/tropej/fmr032. Epub 2011 Apr 20. PMID 21508082
- [Background] Suputtamongkol Y, Hall AJ, Dance DA, Chaowagul W, Rajchanuvong A, Smith MD, White NJ. The epidemiology of melioidosis in Ubon Ratchatani, northeast Thailand. Int J Epidemiol. 1994 Oct;23(5):1082-90. doi: 10.1093/ije/23.5.1082. PMID 7860160
- [Background] Limmathurotsakul D, Wongratanacheewin S, Teerawattanasook N, Wongsuvan G, Chaisuksant S, Chetchotisakd P, Chaowagul W, Day NP, Peacock SJ. Increasing incidence of human melioidosis in Northeast Thailand. Am J Trop Med Hyg. 2010 Jun;82(6):1113-7. doi: 10.4269/ajtmh.2010.10-0038. PMID 20519609
- [Background] Fowler VG Jr, Olsen MK, Corey GR, Woods CW, Cabell CH, Reller LB, Cheng AC, Dudley T, Oddone EZ. Clinical identifiers of complicated Staphylococcus aureus bacteremia. Arch Intern Med. 2003 Sep 22;163(17):2066-72. doi: 10.1001/archinte.163.17.2066. PMID 14504120
- [Background] West TE, Chantratita N, Chierakul W, Limmathurotsakul D, Wuthiekanun V, Myers ND, Emond MJ, Wurfel MM, Hawn TR, Peacock SJ, Skerrett SJ. Impaired TLR5 functionality is associated with survival in melioidosis. J Immunol. 2013 Apr 1;190(7):3373-9. doi: 10.4049/jimmunol.1202974. Epub 2013 Feb 27. PMID 23447684
- [Derived] Booraphun S, Hantrakun V, Siriboon S, Boonsri C, Poomthong P, Singkaew BO, Wasombat O, Chamnan P, Champunot R, Rudd K, Day NPJ, Dondorp AM, Teparrukkul P, West TE, Limmathurotsakul D. Effectiveness of a sepsis programme in a resource-limited setting: a retrospective analysis of data of a prospective observational study (Ubon-sepsis). BMJ Open. 2021 Feb 18;11(2):e041022. doi: 10.1136/bmjopen-2020-041022. PMID 33602702
- [Derived] Wright SW, Lovelace-Macon L, Hantrakun V, Rudd KE, Teparrukkul P, Kosamo S, Liles WC, Limmathurotsakul D, West TE. sTREM-1 predicts mortality in hospitalized patients with infection in a tropical, middle-income country. BMC Med. 2020 Jul 1;18(1):159. doi: 10.1186/s12916-020-01627-5. PMID 32605575
- [Derived] Rudd KE, Hantrakun V, Somayaji R, Booraphun S, Boonsri C, Fitzpatrick AL, Day NPJ, Teparrukkul P, Limmathurotsakul D, West TE. Early management of sepsis in medical patients in rural Thailand: a single-center prospective observational study. J Intensive Care. 2019 Dec 2;7:55. doi: 10.1186/s40560-019-0407-z. eCollection 2019. PMID 31827803
- [Derived] Hantrakun V, Somayaji R, Teparrukkul P, Boonsri C, Rudd K, Day NPJ, West TE, Limmathurotsakul D. Clinical epidemiology and outcomes of community acquired infection and sepsis among hospitalized patients in a resource limited setting in Northeast Thailand: A prospective observational study (Ubon-sepsis). PLoS One. 2018 Sep 26;13(9):e0204509. doi: 10.1371/journal.pone.0204509. eCollection 2018. PMID 30256845